CLINICAL TRIAL: NCT06692738
Title: A Phase III, Randomized, Double-blind, Multicenter, Global Study of Rilvegostomig or Pembrolizumab in Combination With Platinum-based Chemotherapy for the First-line Treatment of Patients With Metastatic Squamous Non-small Cell Lung Cancer Whose Tumors Express PD-L1 (ARTEMIDE-Lung02)
Brief Title: A Global Phase III Study of Rilvegostomig or Pembrolizumab Plus Chemotherapy for First-Line Treatment of Metastatic Squamous Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D702BC00001; 2024-514281-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-10-04; First posted 2024-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ARTEMIDE-Lung02; Rilvegostomig (AZD2936); Non-small cell lung cancer (NSCLC); Bi-specific antibody; T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domain (TIGIT); Programmed death-ligand 1 (PD-L1); Pembrolizumab; Carboplatin; Paclitaxel; Nab-paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Arm A: Rilvegostomig in combination with carboplatin and paclitaxel or nab-paclitaxel followed by rilvegostomig
  Arm B: Pembrolizumab in combination with carboplatin and paclitaxel or nab-paclitaxel followed by pembrolizumab
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Rilvegostomig in combination with carboplatin and paclitaxel or nab-paclitaxel followed by rilvegostomig
  Interventions: Drug: Rilvegostomig; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm B (Active Comparator): Pembrolizumab in combination with carboplatin and paclitaxel or nab-paclitaxel followed by pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Rilvegostomig — Administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: AZD2936
  Arms: Arm A
Drug: Pembrolizumab — Administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: Keytruda
  Arms: Arm B
Drug: Carboplatin — Administered intravenously (IV) on Day 1 of each 21-day cycle up to 4 cycles
Drug: Paclitaxel — Administered intravenously (IV) on Day 1 of each 21-day cycle up to 4 cycles
Drug: Nab-paclitaxel — Administered intravenously (IV) on Days 1, 8, and 15 of each 21-day cycle up to 4 cycles

SUMMARY:
The purpose of ARTEMIDE-Lung02 is to assess the efficacy and safety of rilvegostomig in combination with platinum-based chemotherapy for the first-line (1L) treatment of patients with metastatic squamous non-small cell lung cancer (mNSCLC) whose tumors express programmed death-ligand 1 (PD-L1).

DETAILED DESCRIPTION:
This is a Phase III, two-arm, randomized, double-blind, global, multicenter study assessing the efficacy and safety of rilvegostomig compared to pembrolizumab, both in combination with platinum-based doublet chemotherapy, as a first-line (1L) treatment for patients with squamous metastatic non-small cell lung cancer (mNSCLC) whose tumors express PD-L1 (tumor cells (TC) ≥ 1%).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented squamous NSCLC.
* Stage IV mNSCLC (based on the American Joint Committee on Cancer Edition 8) not amenable to curative treatment.
* Absence of documented tumor genomic mutation results from tests conducted as part of standard local practice in any actionable driver oncogenes for which there are locally approved targeted 1L therapies.
* Provision of acceptable tumor sample to confirm tumor PD-L1 expression TC ≥ 1%.
* At least one lesion not previously irradiated that qualifies as a RECIST 1.1 TL at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with CT or MRI and is suitable for accurate repeated measurements.
* Adequate organ and bone marrow function.

Exclusion Criteria:

* Presence of small cell and neuroendocrine histology components.
* Brain metastases unless asymptomatic, stable, and not requiring steroids or anticonvulsants for at least 7 days prior to randomization. A minimum of 2 weeks must have elapsed between the end of local therapy (brain radiotherapy or surgery) and randomization. Participants must have recovered from the acute toxic effect of radiotherapy (eg, dizziness and signs of increased intracranial pressure) or surgery prior to randomization.
* Any prior systemic therapy received for advanced or mNSCLC.
* Any prior treatment with an anti-PD-1 or anti-PD-L1 agent.
* Any prior exposure to an anti-TIGIT therapy or any other anticancer therapy targeting immune-regulatory receptors or mechanisms.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* Active primary immunodeficiency/active infectious disease(s).
* Active tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2029-02-05 (Estimated); Study Completion 2029-10-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Progression-free survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) or death due to any cause (in the absence of progression).

SECONDARY OUTCOMES:
Landmark overall survival (OS) rates | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Landmark progression-free survival (PFS) rates | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) or death due to any cause (in the absence of progression).
Time to second progression or death (PFS2) | Up to approximately 5 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial progression event), after the start of the first subsequent therapy, or death from any cause, whichever occurs first. The date of the second progression will be recorded by the investigator in the electronic Case Report Form (eCRF) and defined according to local standard clinical practice.
Overall response rate (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants who have a confirmed complete response (CR) or confirmed partial response (PR), by using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
Duration of response (DoR) | Up to approximately 5 years
  DoR is defined as the time from the date of first documented response until the date of documented progression using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) or death due to any cause (in the absence of progression).
Pharmacokinetic (PK) of rilvegostomig | Up to approximately 5 years
  Concentration of rilvegostomig in serum.
Immunogenicity of rilvegostomig | Up to approximately 5 years
  Presence of antidrug antibodies (ADAs), titer, and neutralizing antibodies for rilvegostomig.
Patient-reported physical functioning | Up to approximately 5 years
  Proportion of participants with maintained or improved physical functioning as measured by Patient-Reported Outcomes Measurement Information System Physical Function - Short Form 8c - 7 day (PROMIS PF-SF 8c - 7 day) at each time point.
Patient-reported global health status (GHS)/quality of life (QoL) | Up to approximately 5 years
  Time to deterioration (TTD) of GHS/QoL as measured by the European Organization for Research and Treatment of Cancer Item Library 172 (EORTC IL172). TTD is defined as time from randomization to the date of first deterioration. Deterioration is defined as a worsening change from baseline that reaches a clinically meaningful change threshold.
Patient-reported lung cancer symptoms of non-small cell lung cancer (NSCLC) | Up to approximately 5 years
  Time to deterioration (TTD) in pulmonary symptoms as measured by the Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ).
  TTD is defined as time from randomization to the date of first deterioration.

CONTACTS AND LOCATIONS:
Locations (257):
- United States (68):
  - Research Site, Tucson, Arizona
  - Research Site, Springdale, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Loma Linda, California
  - Research Site, Los Alamitos, California
  - Research Site, Redlands, California
  - Research Site, San Francisco, California
  - Research Site, Walnut Creek, California
  - Research Site, West Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Bay Pines, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Waterloo, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, South Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Camden, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, East Syracuse, New York
  - Research Site, Westbury, New York
  - Research Site, Grand Forks, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Seattle, Washington
  - Research Site, Silverdale, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Plata
  - Research Site, Pilar
  - Research Site, Rosario
- Australia (4):
  - Research Site, Darlinghurst
  - Research Site, Hyde Park
  - Research Site, Southport
  - Research Site, Wollongong
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Krems
  - Research Site, Rankweil
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Kortrijk
  - Research Site, Ottignies
  - Research Site, Sint-Niklaas
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Ijuí
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Taubaté
- Canada (5):
  - Research Site, Saint John, New Brunswick
  - Research Site, Sydney, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Montreal, Quebec
- China (28):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yangzhou
  - Research Site, Yueyang
  - Research Site, Zhengzhou
- France (8):
  - Research Site, Avignon
  - Research Site, La Rochelle
  - Research Site, Lyon
  - Research Site, Nîmes
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Toulon
- Germany (21):
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Gauting
  - Research Site, Giessen
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Homburg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Krefeld
  - Research Site, Minden
  - Research Site, Moers
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Würzburg
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- India (10):
  - Research Site, Calicut
  - Research Site, Delhi
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Puducherry
  - Research Site, Surat
  - Research Site, Varanasi
- Italy (6):
  - Research Site, Florence
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Peschiera del Garda
  - Research Site, Roma
- Japan (21):
  - Research Site, Amagasaki-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kawagoe-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Matsusaka-shi
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Saitama-shi
  - Research Site, Sakai
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Takaoka-shi
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
- Netherlands (6):
  - Research Site, Alkmaar
  - Research Site, Ede
  - Research Site, Groningen
  - Research Site, Leidschendam
  - Research Site, Veldhoven
  - Research Site, Zwolle
- Research Site, Lima, Peru
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Biała Podlaska
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Nakhon Ratchasima
  - Research Site, Songkhla
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Yenimahalle
- United Kingdom (9):
  - Research Site, Aberdeen
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Greater London
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Preston
- Vietnam (4):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca (AZ) group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for Important Protocol Deviation (IPD), but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations (EFPIA)/Pharmaceutical Research and Manufacturers of America (PhRMA) Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/